CLINICAL TRIAL: NCT03630536
Title: TFE Renal Cell Carcinoma: A Prospective Registry and Translational Research Initiative
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: TRRI-REGISTRY
Record Dates: First submitted 2018-06-22; First posted 2018-08-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are limited data regarding the biology and treatment of TFE Renal Cell Carcinoma (TFE RCC). This project provides the infrastructure for acquisition of biological specimens, imaging, and correlative clinical data to facilitate biology studies and characterization of TFE RCC. This registry will collect clinical, demographic, and pathological data, specimens (as available) and imaging from patients with TFE RCC, prospectively. Cases are identified through:

1. Existing clinical and/or cancer registry databases
2. Referrals from clinicians, surgeons, or pathologists
3. Families initiating contact with Registry staff directly

DETAILED DESCRIPTION:
The following data/materials will be collected for this registry study:

Clinical Data: Demographic data, date of diagnosis, pathology, radiological imaging at diagnosis and relapse, signs and symptoms at diagnosis, molecular and biological data, staging details including sites of disease, detailed treatment data (e.g. types and dates of surgeries/interventional therapy (if any), medical/systemic therapy, radiotherapy), response to treatment, dates of progression, types of progression (local or metastatic), and follow-up data. The demographic and clinical data collected are abstracted and entered into an electronic data system secured by password protection (see section 4.3.3). Collection of existing molecular and/or genomic data or analysis that has been performed will also be included.

Research Specimens:

Tissue (fresh/frozen/FFPE) will be requested for all enrolled patients and sent for central review to study pathologist. Then tissue will be stored at CCHMC and future research testing may be conducted on this tissue.

Optional research specimens:

Pending consent specification of family/patient, and resources, specimens may be sent directly to collaborating laboratories to proceed with tumor modeling and drug testing, or other translational research with PI or designee via an IRB approved project.

* Tumor Modeling (Fresh, frozen,): Prospectively collect or retain left-over tumor tissue samples and normal tissue (background kidney) as available, for research purposes.
* Blood: prospectively collected at time of enrollment and at time of relapse
* Urine: prospectively collected at time of enrollment and at time of relapse
* Saliva: prospectively collected at time of or at one time point after at time of enrollment and at time of relapse

Registry clinical data will be correlated with biological/bioinformatic and genomic data. Data stored in the Registry may be used to provide statistical data for scientific presentations and for preparation of peer-reviewed manuscripts. For such purposes all data will be de-identified. Beyond tumor model development and new agent drug testing (if selected in the consent process), data and specimens will be released for IRB approved research proposals upon approval from the TFE RCC Steering Committee.

ELIGIBILITY:
Inclusion Criteria:

* All patients of any age with a suspected diagnosis or confirmed diagnosis of a TFE Renal Cell Carcinoma.
* Unless the patient is deceased, all patients and/or one parent or legal guardian must provide written informed consent as well as HIPAA/release of information consent.

Exclusion Criteria:

* Any patient that has not been diagnosed with TFE Renal Cell Carcinoma

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any age population with a diagnosis of a TFE Renal Cell Carcinoma
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Improving Future Research | From enrollment until data analysis is complete - assessed up to 40 years
  Improving future research by releasing tumor tissue for tumor modeling and drug testing, tumor biology insights, and clinical insights ultimately leading to the development of more effective therapies for children with TFE RCC.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Somers, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States